CLINICAL TRIAL: NCT03445520
Title: Building Better Bridges School Transitions RCT
Brief Title: Building Better Bridges Randomized Control Trial
Acronym: (AIR-B3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Collaborators: University of Rochester (Other); University of Pennsylvania (Other); University of California, Davis (Other); Drexel University (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor/PhD, Health Resources and Services Administration (HRSA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-001459
Record Dates: First submitted 2018-01-15; First posted 2018-02-26 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Transitions; Passport; Building Better Bridges; Snapshot
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition Passport Comparison Group (No Intervention): This group will only receive the Transition Passport, which includes the Transition Checklist, Student Snapshot, Parent/Caregiver Guide, and Student Guide.
- Intervention Coaching Group (Experimental): This group will also receive the Transition Passport, which includes the Transition Checklist, Student Snapshot, Parent/Caregiver Guide, and Student Guide. This group will also receive coaching support to implement these resources. The coach will be a member of the research team who will introduce the resources to the family, briefly teach them fundamental information about the transition process, provide brief coaching phone calls, and help parents identify an appropriate person at the school or district who can work with them to complete the Student Snapshot. This group will also use ParentSquare to enhance and encourage communication between parent and members of the child's school team.
  Interventions: Behavioral: Intervention Coaching Group

INTERVENTIONS:
Behavioral: Intervention Coaching Group — Parents in this group receive six, 1 hour, coaching sessions with a research staff coach, to discuss key information about transitions (knowing parent's rights about special education services, communicating effectively with school staff, knowing the roles of the school team members, how to develop and share your Snapshot, and what to do with your child over the summer to help with the transition). The coach will encourage the parent to identify a school staff member to help with preparing for the transition. If the post transition school team is not able to participate in a pre-transition meeting, then the coach will encourage the parent to share the Student Snapshot with the post-transition teacher(s) and school team when the new school year begins in the Fall.
  Arms: Intervention Coaching Group

SUMMARY:
In this study, the investigators will randomize 20 families per site (across 4 sites) to be in the BBB Transition Passport Only Group or BBB Intervention Group. Both groups will receive the BBB Transition Passport, which include the Transition Checklist, Student Snapshot, Parent/Caregiver Guide, and Student Guide. In addition to receiving the Transition Passport, the BBB Intervention Group will also receive coaching support to implement these resources. This coaching will include a member of the research team assigned as a coach for each family. This coach will introduce the resources to the family, briefly teach them fundamental information about the transition process, provide brief coaching phone calls, and guide parents in using the tools and requesting help from the child's provider(s).

The investigators will be testing the differences between these two groups in terms of: 1) quality of the transition as reported by the parent and teacher, 2) self-efficacy of the parent during the transition process, 3) child school engagement and behavior during the transition as rated by the teacher and parent, and 4) the quality of the child's team to communicate about information important to the child's transition.

DETAILED DESCRIPTION:
Building Better Bridges (BBB), will evaluate an intervention designed to support the needs of students with autism who are transitioning from either preschool to elementary school, or from elementary to secondary school. In this randomized controlled trial, the investigators will randomly assign a total of 160 families (40 families/site, across 4 sites, over 2 years) to one of two intervention groups: BBB Transition Passport Only Group (Comparison) or BBB Intervention Group. Both groups will receive the BBB Transition Passport, which include the Transition Checklist, Student Snapshot, Parent/Caregiver Guide, and Student Guide. In addition to receiving the Transition Passport, the BBB Intervention Group will also receive coaching support to implement these resources. The coach will be a member of the research team who will introduce the resources to the family, briefly teach them fundamental information about the transition process, provide brief coaching phone calls, and help parents identify an appropriate person at the school or district who can work with them to complete the Student Snapshot.

The research staff will first recruit interested schools, and school administrators will identify potential teachers who may have eligible students. If the teacher agrees to participate, he/she will send the study flyer home to parents where parents can either call the study phone line to learn more, or can fill out the study interest portion of the flyer and turn it in to their teachers. Parents who fill out the interest sheet will be contacted by the research staff. Interested parents can also contact research staff. All parents will receive a screening over the telephone to determine eligibility, which will include an Social Communication Questionnaire (SCQ) over the phone and will ask if their child has received a diagnosis of Autism by the administration of an Autism Diagnostic Observation Schedule (ADOS) or any other official diagnosis. The investigators will accept an ADOS diagnosis within one year for children in preschool and within three years for students transitioning to secondary school.. If an ADOS or any record of an official diagnosis is not provided, the research staff will schedule a time to administer the ADOS to determine eligibility. We will also ask if the child has a record of a cognitive test like the Stanford Binet-5. If parents do not have a record or if it has been over a year since the pre-school child or over 3 years since the older child has had one, the research staff will also schedule with the parents to administer it around the same time as the ADOS.

After the initial phone screen and verification of autism diagnosis, the parent will be consented and then will complete baseline T1 measures. Pre-transition teachers will complete T1 measures as well. Schedule of measures can be found in the Outcome Measures Section.

Following enrollment into the study, the child will be randomized to one of two treatment groups, BBB Comparison Group(Control) or BBB Intervention Group.

Families randomized to the control group will only have access to the BBB Transition Passport, which consists of the Transition Checklist, Parent Guide, Student Guide, and the Student Snapshot. A hard copy of these tools will be given to them. We will also provide them with a link to download them online through LiveBinder (online website).

Families randomized to the BBB Intervention group will be enrolled in ParentSquare if they agreed to it in the consent form. ParentSquare is an app that provides a safe and secure platform for program-to-parent communication. ParentSquare is in compliance with Family Educational Rights and Privacy Act (FERPA). Any school team members who want to use ParentSquare will be consented to use it and agree to allow the de-identified data from ParentSquare to be used for research purposes. The participants in this group will also have access to download the tools and share them with each other.

Parents in the intervention group will also receive six, 1 hour, coaching sessions (one session per month for six months), with a research staff coach, to discuss key information about transitions (knowing parent's rights about special education services, communicating effectively with school staff, knowing the roles of the school team members, preparing their child over the summer, developing and sharing their Snapshot). These coaching sessions will occur individually (in-person or by telephone) during the pre-transition school year.

In addition, parents will receive ongoing 1-2 monthly follow up phone calls (10 minutes each) to see how the transition planning is going, to help the parent problem-solve around any concerns about the transition, and to encourage the parent to implement all components of the intervention (including conducting at least one school visit, working on the student guide, and completing the Student Snapshot with the school team). These coaching calls are expected to start in February during the pre-transition school year and continue through November of the post-transition year. Coaching calls are designed to be flexible and brief and can occur in person or by telephone, or by a secure internet-based platform (Zoom), depending on the parent's preference.

The coach will encourage the parent to identify a school staff member to help with preparing for the transition. This person can be the child's teacher, provider, or someone else from the school or district who can assist with the child's transition. The coach will encourage the parent to work with this school person to arrange a meeting prior to the transition (or join an existing meeting), for the purpose of completing the Student Snapshot and meeting with a post-transition teacher or staff from the receiving school, if possible. This school staff person can also help to recruit other school team members working on the transition process and to utilize Parent Square for all communication and sharing of transition materials. Any team member involved in the transition will be offered to be consented and given access to Parent Square. This meeting will occur at a time convenient for the school team, likely in April or May. If the post-transition school personnel can attend the meeting (if known prior to the transition), they will also be consented for the study form. During this meeting, everyone will work together to complete the BBB Passport materials.

If the post transition school team is not able to participate in a pre-transition meeting, then the coach will encourage the parent to share the Student Snapshot with the post-transition teacher(s) and school team when the new school year begins in the Fall.

ELIGIBILITY:
Inclusion Criteria:

* Children:

  * Transitioning into kindergarten or secondary school (middle/high school)
  * Parent-rated SCQ total score > 15 and AT LEAST one of the following:

    * Positive ADOS-2 administered by research-reliable study personnel
    * Expert medical diagnosis or educational classification of ASD
  * Under-resourced, defined by:

    * Attending or transitioning into a Title I school (a school that receives federal funding to improve the performance of economically disadvantaged students)or rural school
    * Family income is under 250% of the federal guidelines for poverty rate (i.e., meets federal requirements to qualify for free or reduced lunch)
  * Parent/Caregiver willing to participate

(Site PIs may request eligibility review by PIs across all AIR-B sites if a school is not Title I or rural but is demonstrably low-resource)

Adults:

* Must be a parent/caregiver of a child who meets criteria above
* Must be a provider/teacher/school administrator or other adult involved in either the pre-transition process or the post transition process for a participating child.

Exclusion Criteria:

* Children:

  * Not transitioning into kindergarten or secondary school
  * No ASD diagnosis
  * Not meeting study criteria for classification as under-resourced
  * Parent/Caregiver unwilling to participate

Adults:

* Not a parent/guardian of a child with ASD
* Not part of a participating child with ASD's pre or post transition team

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Transition Evaluation Questionnaire (TEQ) | entry (1st month of the study)
  This measure was created by the research team. We capture the parents and pre and post transition personnels thoughts on how the transition process is going for the child at the beginning of the study and throughout the big school transition. Communication and transition planning at home and school is also captured in this measure. It is rated from 0(not knowing anyone in the child's school) to 5 (very satisfied, very effective, high support) with the child's transition process. We expect to start around 1(not effective/no communication) or 2 (little effective/little successful) at the beginning of the study and end at a 4 (mostly successful/effective) or a 5(very satisfied/effective).
Transition Evaluation Questionnaire (TEQ) | end of school year (4th month of the study)
  This measure was created by the research team. We capture the parents and pre and post transition personnels thoughts on how the transition process is going for the child at the beginning of the study and throughout the big school transition. Communication and transition planning at home and school is also captured in this measure. It is rated from 0(not knowing anyone in the child's school) to 5 (very satisfied, very effective, high support) with the child's transition process. We expect to start around 1(not effective/no communication) or 2 (little effective/little successful) at the beginning of the study and end at a 4 (mostly successful/effective) or a 5(very satisfied/effective).
Transition Evaluation Questionnaire (TEQ) | 6 weeks post new school year (7th month of the study)
  This measure was created by the research team. We capture the parents and pre and post transition personnels thoughts on how the transition process is going for the child at the beginning of the study and throughout the big school transition. Communication and transition planning at home and school is also captured in this measure. It is rated from 0(not knowing anyone in the child's school) to 5 (very satisfied, very effective, high support) with the child's transition process. We expect to start around 1(not effective/no communication) or 2 (little effective/little successful) at the beginning of the study and end at a 4 (mostly successful/effective) or a 5(very satisfied/effective).
Transition Evaluation Questionnaire (TEQ) | 3 months post new school year (10th month of the study)
  This measure was created by the research team. We capture the parents and pre and post transition personnels thoughts on how the transition process is going for the child at the beginning of the study and throughout the big school transition. Communication and transition planning at home and school is also captured in this measure. It is rated from 0(not knowing anyone in the child's school) to 5 (very satisfied, very effective, high support) with the child's transition process. We expect to start around 1(not effective/no communication) or 2 (little effective/little successful) at the beginning of the study and end at a 4 (mostly successful/effective) or a 5(very satisfied/effective).

SECONDARY OUTCOMES:
Engagement vs.Disaffection | entry (1st month of the study), end of school year (4th month of the study), 6 weeks post new school year (7th month of the study), and 3 months post new school year (10th month of the study)
  This measure will provide information on the change of each child's behavior throughout the transition process. It will be measure through the parents and school personnels perspectives. Filled out by parents and school personnel.
Social Dynamics of Intervention_ASD (Autism Spectrum Disorder)- SoDI | entry (1st month of the study), end of school year (4th month of the study), 6 weeks post new school year (7th month of the study), and 3 months post new school year (10th month of the study)
  This measure shows the level of support and how well connected parents and school personnel of the children in the study are in their community and in their child's school setting. Filled out by parents and school personnel.
Parent Engagement (ESE) | entry (1st month of the study), end of school year (4th month of the study), 6 weeks post new school year (7th month of the study), and 3 months post new school year (10th month of the study)
  This measure will demonstrate each parent's knowledge and engagement in their child's transition process.
Community Capital | entry and 3 months post transition (10th month of the study)
  This survey measures how each parent's community involvement/importance influences their behavior.
Usability & Acceptability Form | Parents: end of school year (4th month of the study), 6 weeks post-transition (7th month of the study), 3 months post-transition(10th month of the study) Pre-transition personnel: 4th month of study Post transition personnel: 10th month of study
  Measures how useful each tool and component of the intervention was for parents and school personnel.
Strategies Survey | Parents: end of school year (4th month of study), 6 weeks post-transition(7th month of study) Pre-transition personnel: entry and end of school year (4th month of study) Post-transition personnel: 7th month of study, 10th month of study
  Description of strategies that help the child with the transition process and schooling in general.
Transition Practices | Pre-transition personnel: at entry Post-transition personnel: 6 weeks post-transition(7th month of the study)
  Measures each school personnel's level of engagement that helps with the transition process, such as what tools, activities, and strategies they used to help the child.
Burnout Measure | Pre-transition personnel: entry Post-transition personnel: 6 weeks post-transition(7th month of study)
  Measures each school personnel's burnout level at entry.
School Situations Questionnaire (SSQ) | Pre-transition personnel: entry, end of school year (4th month of study) Post-transition personnel: 6 weeks post-transition (7th month of study) and 3 months post-transition(10th month of study)
  Describes child's behavior in different school situations and the severity of the behavior.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UC Davis, Davis, California
  - University of Rochester, Rochester, New York
  - UPENN, Philadelphia, Pennsylvania